CLINICAL TRIAL: NCT04006730
Title: Analysis of the Pharmaceutical Validation of Picc Line Installation Requests at the Nîmes University Hospital
Acronym: PICCLINIC
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Other Study IDs: Local/2018/VC-01
Record Dates: First submitted 2019-07-01; First posted 2019-07-05 (Actual); Last update posted 2024-01-26 (Actual); Status verified 2019-06

CONDITIONS: Parenteral Nutrition
MeSH Terms: conditions — Hyperphagia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The picc line is a central venous catheter inserted peripherally into a deep vein in the arm (cephalic, basilic or axillary) whose distal end is located at the junction of the superior vena cava / atrium.

It is installed for a minimum of 7 days (1), and can be stored for up to 6 months or more if it is functional. For treatments with an indication of more than 3 months, it is common practice to place an implantable catheter chamber. The main indications for picc line placement are: long-term antibiotic therapy, parenteral nutrition, chemotherapy or long-term venous approach when difficulties are encountered in applying a peripheral venous route to the patient.

Quickly adopted by medical teams, picc lines are not without risk, however, and three complications are mainly reported: catheter obstruction, deep vein thrombosis and infections.

In order to avoid any risk of unnecessary complications, it therefore seems appropriate to target the most appropriate device upstream of the procedure according to the provisional indication.

An inventory of pharmaceutical interventions carried out during picc line requests would make it possible to lay the foundations for considering actions to be implemented with the various services requesting picc line and proposals for improvement for the follow-up of patients with picc line to reduce the risk of complications.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged 18 or over, hospitalized at the University Hospital of Nîmes
* Benefiting from a pharmaceutical validation of the demand for picc line connected

Exclusion Criteria:

* The patient is opposed to participating in this study

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patients included in the study are patients aged at least 18 years old, hospitalized at the University Hospital of Nîmes and benefit from a pharmaceutical validation of the connected request for picc line in the Xplore® software.
Sampling Method: Non-Probability Sample
Enrollment: 277 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2019-03-14 (Actual); Study Completion 2019-03-14 (Actual)

PRIMARY OUTCOMES:
estimate the prevalence of requesting pharmaceutical interventions with a criticality greater than or equal to 2 accepted. | 2018

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Nimes, Nîmes, France

REFERENCES:
- [Derived] Chasseigne V, Buisson M, Serrand C, Leguelinel-Blache G, Kinowski JM, Goupil J, Beregi JP, Frandon J. Pharmaceutical Analysis of Peripherally Inserted Central Catheter Requests Increases the Use of Single-Lumen Catheters: A Prospective Pilot Study. J Patient Saf. 2022 Dec 1;18(8):e1238-e1242. doi: 10.1097/PTS.0000000000001065. Epub 2022 Aug 2. PMID 35858479
- [Derived] Buisson M, Leguelinel G, Bastide S, Beregi JP, Kinowski JM, Frandon J, Chasseigne V. A new clinical approach to improve the appropriate use of peripherally inserted central catheters: a prospective study. Eur J Hosp Pharm. 2021 Nov;28(Suppl 2):e134-e139. doi: 10.1136/ejhpharm-2020-002483. Epub 2021 Jan 7. PMID 33414259